CLINICAL TRIAL: NCT00569413
Title: A Combined Psycho-pharmacological and Brain Imaging Study of Human Sexuality
Status: Suspended | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Prof. Roland Chisin, Hadassah Medical Organization
Other Study IDs: 281207HMO-CTIL; First 978[1].07
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Hypoactive Sexual Desire Disorder; Erectile Dysfunction
Keywords: Sex; brain imaging; dopamine; sexual disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Erectile Dysfunction; Coitus; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Healthy control subjects (n=20) age 21-65 who do not suffer from a psychiatric diagnosis or neurological damage, are under age, or are pregnant women
- 2: 20 patients who suffer from sexual disorder (reduced sexual desire or sexual function) from a sexual disorder clinic, age 21-65, without any other psychiatric disorder, neurological damage, are not under age or pregnant women.

SUMMARY:
The current study combines a molecular genetic perspective, self report and brain imaging to the study of human sexuality in control subjects and individuals from a sexual disorder clinic. The investigators hypothesize that the variability in components of the brain dopaminergic system expressed in the mesolimbic reward system can explain variability in human sexuality, especially in desire and pleasure associated with sex.

DETAILED DESCRIPTION:
We intend to combine molecular genetics of the dopamine receptors (D2, D3 D4 and D5) and brain imaging using 11 C Raclopride in Positron Emission Tomography (PET). 11 C Raclopride is a ligand which binds to the dopamine receptor D2 and can measure dopamine release during pleasure or anticipatory reward associated with sex. The current proposal will measure changes in DRD2 receptor occupancy using 11 C Raclopride following explicit visual sexual desire cues in healthy control subjects and individuals who suffer from sexual dysfunction. This is in order to determine how individual genotypes modulate dopamine release in vivo in the human brain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and patients
* Age 21-65
* Male or female

Exclusion Criteria:

* Psychiatric diagnosis/psychosis
* Neurological damage associated with loss of consciousness
* Infectious disease HIV
* Herpes
* Syphilis
* Hyperactivity treated with ritalin
* Pregnant women
* Under age

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of healthy volunteers from the general public. A group of patients who suffer from sexual disorder from a primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Brain Imaging data of DRD2 receptor occupancy during watching a sex videotape and neutral videotape | 2 Brain imaging sessions a week apart

SECONDARY OUTCOMES:
Questionnaire ratings of human sexuality, pleasure, and anticipatory reward | Taken during brain scans

CONTACTS AND LOCATIONS:
Overall Officials: Aviv M Weinstein, Ph.D, Principal Investigator — Hadasah Medical Organization, Jerusalem Israel